CLINICAL TRIAL: NCT02721550
Title: A Perspective Trial of Sodium Glycididazole Combined With Preoperatie Concurrent Chemoradiotherapy for Locally Advanced Squamous Cell Esophageal Carcinoma
Brief Title: A Trial of CMNa Combined With Preoperatie Concurrent Chemoradiotherapy for Locally Advanced ESCC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The number of enrollment cases is too small.
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, president, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMNAER1
Record Dates: First submitted 2016-03-09; First posted 2016-03-29 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — sodium glycididazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium Glycididazole (Experimental): Sodium Glycididazole：800mg/m2，finished in 30 minutes,within 60 minutes after intravenous drip for radiation therapy.Three times a week (once every other one day),before radiation therapy. Chemotherapy Paclitaxel:45 mg/m²,d1,week 1-4 Cisplatin:20 mg/m²,d1,week 1-4 OR Docetaxel: 75 mg / m², 1 day or divided into D1, D8 days, 21 days / cycle. Cisplatin: 75 mg / m², divided into D1-D3 days or D1-D5 days, 21 days / cycle. Or nedaplatin: 80 mg / m², 21 days / cycle.
  OR 5-FU: 500 mg / m² / day, divided into D1 ~ D5 for use, 21 days / cycle. Cisplatin: 75 mg / m² / day, divided into D1-D3 day or D1-D5 days, 21 days / cycle. Or nedaplatin: 80 mg / m², 21 days / cycle 3DCRT/IMRT:2.0Gy/f/day,T40Gy/20f,week 1-4
  Interventions: Drug: Sodium Glycididazole

INTERVENTIONS:
Drug: Sodium Glycididazole — 800mg/m2，dissolved in 100ml physiological saline(Now with chef),ivgtt,finished in 30 minutes,within 60 minutes after intravenous drip for radiation therapy.Three times a week (once every other one day),before radiation therapy, total 4 weeks course.

SUMMARY:
This is a perspective, multicenter,single arm, open label study to evaluate the efficacy and safety of treatment with CMNa combined with preoperatie concurrent chemoradiotherapy in patients with locally advanced squamous cell esophageal carcinoma . Analyses of primary objective (pathologic Complete Response) will be done as defined in the protocol.

DETAILED DESCRIPTION:
The primary end ponit of this study is pathological complete response.And the primary hypothesis is the CMNa will improve patholofical response rate and thus improve OS、DFS. Assuming bilateral a=0.05, statistical power of 80%.The total sample size is 40 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to study entry
2. Patients with ESCC in thoracic segment which is resectable（T2-3，N0-1，M0） confirmed by imaging and pathology or cytology;
3. Patients have tumor lesions which can be objectively measured ,the length of tumor:≤8cm, the width of tumor:≤5cm;If the tumor cross the GEJ and violate the proximal stomach, the tumor must include esophagus and GEJ. The tumor is less than 2cm of the stomach
4. Not infringe bronchial wall; no esophagus-tracheal fistula.
5. normal bone marrow reserve: ANCcount ≥1500/mm3;platelet count ≥100,000/mm3,hemoglobin≥9g/dl
6. normal hepatic funcion:bilirubin level ≤1.5×ULN;AST/ALT≤1.5×ULN
7. normal renal function: serum creatinine≤1.5mg/dl and calculated creatinine clearance ≥60ml/min
8. normal cardiac function
9. ECOG PS of 0 or 1
10. Expected lifetime≥3 months
11. Subjects tumor tissue available for the relevant biomarker detection

Exclusion Criteria:

1. Female subject who is during pregnancy or lactation, and the subject who have fertility don't take effective contraception during study.
2. Any mental illness or nervous system lesions or can't tell treatment response clearly (such as cerebrovascular accident sequelae)
3. Any serious uncontrolled disease and infection, such as severe heart, liver, kidney diseases or diabetes, can't complete the treatment plan
4. Patients who have other malignant lesions, except curable skin cancer (non- melanoma skin cancer),carcinoma in situ of cervix or serve disease cured for 5 years
5. Primary lesions were multifocal
6. Patients with distant metastasis. A small amount of stomach tumor violate GEJ or the distal esophageal.
7. Patients who have obvious esophageal ulcers or have above moderate pains in chest-back or have symptoms of esophageal perforation
8. received anti-cancer treatment of esophageal cancer before the group, including surgery, radiotherapy, chemotherapy (induction of chemotherapy before the group is greater than or equal to two cycles).
9. Cervical esophageal cancer confirmed by iconography
10. Not esophageal squamous carcinoma confirmed by pathology or cytology
11. History of active hepatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
pathologic Complete Response | 1 months
  TRG-cited from Mandard AM, Dalibard F, Mandard JC, Marnay J, Henry-Amar M, Petiot JF, Roussel A, Jacob JH, Segol P, Samama G, Pathologic assessment of tumor regression after preoperative chemoradiotherapy of esophageal carcinoma. Cancer, 73, 2680-2686, 1994.

SECONDARY OUTCOMES:
Overall Survival | 36 months
Disease-Free Survival | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, Ph.D, M.D, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (9):
- China (9):
  - Qianfoshan Hospital of Shandong, Jinan, Shandong
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - Jining NO.1 People's Hospital, Jining, Shandong
  - Liaocheng People Hospital, Liaocheng, Shandong
  - Qingdao Center Medical Group, Qingdao, Shandong
  - Rizhao City People 's Hospital, Rizhao, Shandong
  - Fei Cheng People's Hospital, Tai’an, Shandong
  - An Qiu People's Hospital, Weifang, Shandong
  - The Fourth People's Hospitalof Zibo, Zibo, Shandong

IPD SHARING:
Plan to Share IPD: No